CLINICAL TRIAL: NCT04167085
Title: NOrth American Study for the Treatment of Recurrent epIstaxis With DoxycycLine: The NOSTRIL Trial
Acronym: NOSTRIL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Justin McWilliams, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 16-001827
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Results first posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-06

CONDITIONS: Epistaxis
Keywords: Epistaxis; Hereditary Hemorrhagic Telangiectasia; HHT; Doxycycline; Nosebleed
MeSH Terms: conditions — Epistaxis; Telangiectasia, Hereditary Hemorrhagic | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doxycycline, then Placebo (Experimental): Doxycycline for a period of 2 months followed by a 1-month washout period, and then placebo for a further 2 months period followed by a 1-month washout period.
  Interventions: Drug: Doxycycline; Other: Placebo
- Placebo, then Doxycycline (Experimental): Placebo for a period of 2 months followed by a 1-month washout period, and then Doxycycline for a further 2 months period followed by a 1-month washout period.
  Interventions: Drug: Doxycycline; Other: Placebo

INTERVENTIONS:
Drug: Doxycycline — Doxycycline, 100 mg twice a day for 2 months
Other: Placebo — Matching placebo, twice a day for 2 months

SUMMARY:
The purpose of this research study is to determine whether Doxycycline can be used to control nosebleeds (epistaxis) for patients with Hereditary Hemorrhagic Telangiectasia (HHT). Patients with HHT will be randomized to one of 2 study arms: Doxycycline or Placebo for a period of 2 months followed by a 1-month washout period before switching treatments for a further 2 months period. Observation and evaluation will continue for a period of one month after treatment is completed.

DETAILED DESCRIPTION:
This study will analyze the effect of doxycycline on nosebleeds in hereditary hemorrhagic telangiectasia (HHT), a rare and debilitating medical condition. Patients with HHT have a variety of vascular abnormalities, including changes in their nasal vasculature that result in chronic, severe nosebleeds. These nosebleeds have been shown to significantly reduce the quality of life in HHT and can be severe enough to require emergent blood transfusion. Current therapies to control nosebleeds in HHT, which include both medications and surgical treatments, are inconsistently effective and associated with a variety of problematic side effects and complications.

Doxycycline is a common, FDA-approved antibiotic medication that has been used by physicians for decades. It is a safe medication that can be used on an outpatient basis for extended periods of time with minimal side effects. Recent research has shown that doxycycline is a potent inhibitor of angiogenesis, the process of new blood vessel development. Since the vascular abnormalities in HHT form due to uncontrolled angiogenesis, it follows that doxycycline may have potential in treating HHT. A growing body of research demonstrates the efficacy of doxycycline in treating a variety of vascular conditions, including cancer of the breast, duodenum, liver prostate, and lung. Our trial will be the first to analyze the efficacy of doxycycline in treating HHT epistaxis.

This a randomized, double-blind, crossover study design. Each patient will take both placebo and doxycycline. Since this is a cross-over study, half the participants will start out with taking placebo and half start with doxycyline and then switch halfway through. After a baseline observation period, participants will be given doxycycline at 100 mg twice a day, or an identical-appearing placebo, for a period of three months. Each month they will be seen be a physician, who will take a detailed clinical history and perform a physical examination. Further, each month the patient will have blood testing to assess blood loss, and fill out scientifically validated surveys to assess quality of life and the severity of bleeding. Following this three month treatment period, participants will be observed for one additional month, with one additional blood test and clinical assessment performed after this month.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of definite HHT by the Curacao criteria or genetic diagnosis of HHT
* Epistaxis severity during observation month at least moderate by Epistaxis Severity Score (ESS) evaluation
* For female participants, a negative pregnancy test at Day -1 and agree to use birth control during treatment and for 28 days following cessation of Doxycycline

Exclusion Criteria:

* Use of medication(s) contraindicated with doxycycline use within 14 days prior to the study (including barbiturates, tegretol, dilantin, warfarin, isotretinoin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- 100 UCLA Medical Plaza, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | Doxycycline, Then Placebo | Placebo, Then Doxycycline
Started | 13 | 13
Day 1 | 12 | 12
Completed | 11 | 12
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1
Period: First Intervention (2 Months)
Arm/Group | Doxycycline, Then Placebo | Placebo, Then Doxycycline
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0
Period: Washout (1 Month)
Arm/Group | Doxycycline, Then Placebo | Placebo, Then Doxycycline
Started | 11 | 12
Completed | 10 | 12
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention (2 Months)
Arm/Group | Doxycycline, Then Placebo | Placebo, Then Doxycycline
Started | 10 | 12
Completed | 10 | 12
Not Completed | 0 | 0
Period: Washout (1 Month)
Arm/Group | Doxycycline, Then Placebo | Placebo, Then Doxycycline
Started | 10 | 12
Completed | 10 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxycycline, Then Placebo | Placebo, Then Doxycycline | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (12.9) | 63.6 (13.8) | 57.4 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 9 | 15
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26
Epistaxis Severity Scale (ESS) score [Mean (Standard Deviation); unit: Score on a scale] — Epistaxis Severity Scale (ESS) for Hereditary Hemorrhagic Telangiectasia, is based on 6 nosebleed variables such as frequency and duration which are reported by patients.The ESS has a minimum value of 0 and maximum value of 10, with 10 representing more severe epistaxis.
  Score on a scale | 6.3 (1.2) | 5.7 (1.5) | 6.0 (1.4)
Quality of Life [Mean (Standard Deviation); unit: Score on a scale] — The 12-item Short Form (SF-12) is a survey designed for use with patients with multiple chronic conditions. This 12-item scale can be used to assess the physical and mental health of respondents. 10 of the 12 questions are answered on a 5-point Likert scale and 2 are answered on a 3-point Likert scale. The questions are then scored and weighted into 2 subscales, physical health and mental health. Respondents can have a score that ranges from 0-100 with 100 being the best score and indicating high physical or mental health.
  Score on a scale
    SF-12 Physical | 43.6 (10.7) | 40.2 (9.7) | 41.9 (10.2)
    SF-12 Mental | 47.0 (12.5) | 54.4 (6.4) | 50.7 (10.4)
Hemoglobin level [Mean (Standard Deviation); unit: g/dl] | 12.8 (2.5) | 12.3 (2.4) | 12.5 (2.4)
Ferritin Level [Mean (Standard Deviation); unit: ng/ml] | 71.1 (83.7) | 98.1 (186.3) | 85.1 (144.1)
Number of monthly iron infusions [Number; unit: participants]
  No infusions | 9 | 11 | 20
  1 infusion | 2 | 1 | 3
  2 infusions | 1 | 1 | 2
  Not reported | 1 | 0 | 1
Number of monthly blood transfusions [Number; unit: participants]
  0 transfusions | 12 | 12 | 24
  1 transfusion | 0 | 1 | 1
  Not reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Epistaxis
Description: Change in number of bleeding episodes per week by participant self-report via nosebleed diary
Time Frame: Baseline, post-washout - approximately 6 months
Population: All participants who received each intervention and completed all study visits were included in the efficacy analysis
Measure: Mean (Standard Deviation); unit: Nosebleeds per week
Groups:
- Doxycycline: Participants who received Doxycycline, 100 mg twice a day for 2 months in either the first or second intervention period of the study
- Placebo: Participants who received placebo (matching Doxycycline 100mg) twice a day for 2 months in either the first or second intervention period of the study.
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 22 | 22
Nosebleeds per week | -1.68 (6.55) | 1.14 (4.44)
Statistical Analysis 1: Comparison: Doxycycline vs Placebo; Test type: Superiority; p = 0.16, Wilcoxon (Mann-Whitney) — Threshold p<0.0167 - Because 3 primary outcomes were prespecified, the familywise error rate was adjusted for 3 endpoints: 0.05/3

2. Primary Outcome: Duration of Epistaxis
Description: Change in duration of bleeding per week by patient self-report via nosebleed diary
Time Frame: Baseline, post-washout - approximately 6 months
Population: All participants who received each intervention and completed all study visits were included in the efficacy analysis
Measure: Mean (Standard Deviation); unit: Minutes per week
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 22 | 22
Minutes per week | -41.17 (159.26) | 24.36 (58.03)
Statistical Analysis 1: Comparison: Doxycycline vs Placebo; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Change in Severity of Epistaxis
Description: Epistaxis Severity Scale (ESS) for Hereditary Hemorrhagic Telangiectasia, is based on 6 nosebleed variables such as frequency and duration which are reported by patients.The ESS has a minimum value of 0 and maximum value of 10, with 10 representing more severe epistaxis.
Time Frame: Baseline, post-washout - approximately 6-months
Population: All participants who received each intervention and completed all study visits were included in the efficacy analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 22 | 22
score on a scale | -.095 (1.55) | -0.32 (1.3)
Statistical Analysis 1: Comparison: Doxycycline vs Placebo; Test type: Superiority; p = 0.19, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change in Quality of Life
Description: The 12-item Short Form (SF-12) is a survey designed for use with patients with multiple chronic conditions. This 12-item scale can be used to assess the physical and mental health of respondents. 10 of the 12 questions are answered on a 5-point Likert scale and 2 are answered on a 3-point Likert scale. The questions are then scored and weighted into 2 subscales, physical health and mental health. Respondents can have a score that ranges from 0-100 with 100 being the best score and indicating high physical or mental health.
Time Frame: Baseline, post-washout - approximately 6 months
Population: All participants who received each intervention and completed all study visits were included in the efficacy analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 22 | 22
score on a scale
  SF-12 Physical | 2.21 (6.94) | -0.83 (6.72)
  SF-12 Mental | -0.63 (9.97) | -0.63 (9.74)
Statistical Analysis 1: Comparison: Doxycycline vs Placebo; SF-12 Physical; Test type: Superiority; p = 0.24, Wilcoxon (Mann-Whitney) — Threshold p=0.05
Statistical Analysis 2: Comparison: Doxycycline vs Placebo; SF-12 Mental; Test type: Superiority; p = 0.35, Wilcoxon (Mann-Whitney) — Threshold p=0.05

5. Secondary Outcome: Change in Ferritin Level
Time Frame: Baseline, post-washout - approximately 6 months
Population: All participants who received each intervention and completed all study visits were included in the efficacy analysis
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 22 | 22
ng/ml | 14.9 (72.82) | -47.4 (214.83)
Statistical Analysis 1: Comparison: Doxycycline vs Placebo; Test type: Superiority; p = 0.50, Wilcoxon (Mann-Whitney) — Threshold p=0.05

6. Secondary Outcome: Change in Hemoglobin Level
Time Frame: Baseline, post-washout (approximately 6 months)
Population: All participants who received each intervention and completed all study visits were included in the efficacy analysis
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 22 | 22
g/dl | 0.26 (1.09) | -0.12 (1.19)
Statistical Analysis 1: Comparison: Doxycycline vs Placebo; Test type: Superiority; p = 0.30, Wilcoxon (Mann-Whitney) — Threshold p=0.05

7. Secondary Outcome: Change in Monthly Units of Packed Red Blood Cells (PRBCs) Transfused
Time Frame: Baseline, post-washout (approximately 6 months)
Population: All participants who received each intervention and completed all study visits were included in the efficacy analysis
Measure: Mean (Standard Deviation); unit: count of PBRC units
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 22 | 22
count of PBRC units | 0 (0.31) | 0 (0)
Statistical Analysis 1: Comparison: Doxycycline vs Placebo; Test type: Superiority; p = 1.00, Wilcoxon (Mann-Whitney) — Threshold p=0.05

8. Secondary Outcome: Incidence of Treatment Failure
Description: Treatment failure, defined as need for nasal surgery or other epistaxis treatments
Time Frame: Baseline, post-washout (approximately 6 months)
Population: All participants who received each intervention and completed all study visits were included in the efficacy analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 22 | 22
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Baseline, post-washout (approximately 6 months)
Arm/Group | Doxycycline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 6/23 | 6/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxycycline (N=23) | Placebo (N=22)
GI bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) — chronic gastrointestinal bleeding, ongoing since before enrollment
Flu-like symptoms (Infections and infestations) | 0 (0) | 1 (1)
Prolonged nosebleed requiring cauterization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia hospitalization (Infections and infestations) | 0 (0) | 1 (1)
Allergy-like symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat infection (Infections and infestations) | 0 (0) | 1 (1)
Metastatic lung cancer dx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sinus infection (Infections and infestations) | 1 (1) | 0 (0)
Foot infection (Infections and infestations) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Emesis (Gastrointestinal disorders) | 1 (4) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/85/NCT04167085/Prot_SAP_000.pdf